CLINICAL TRIAL: NCT02649257
Title: Influence of an Capsular Tension Ring on the Rotation of an Intraocular Lens (Aspira®-aA Also Known as MC 6125 AS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EK-Nr.: 1435/2014
Record Dates: First submitted 2015-12-22; First posted 2016-01-07 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Cataract
Keywords: IOL rotation; capsular tension ring; IOL rotational stability
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Lenses, Intraocular

ARMS (1):
- MC 6125 AS IOL + CTR (Experimental): All patients received the same procedure: cataract surgery with phakoemulsification, implantation of a capsular tension ring (CTR13/11) and implantation of an intraocular lens (MC 6125 AS).
  Interventions: Procedure: cataract surgery; Device: intraocular lens (MC 6125 AS); Device: capsular tension ring (CTR 13/11)

INTERVENTIONS:
Procedure: cataract surgery
Device: intraocular lens (MC 6125 AS)
Device: capsular tension ring (CTR 13/11)

SUMMARY:
The purpose of this study is to observe the axial IOL rotation after surgery with a capsular tension ring (CTR) and a MC6125 AS IOL.

At the end of surgery the orientation of the IOL is documented with a short video clip via the operating microscope unit. Follow-up examinations are performed 1 hour, 1 week and 6 months after surgery. Rotational stability of the IOL is assessed using retroillumination images with a method to avoid bias from cyclorotation or head tilt.

ELIGIBILITY:
Inclusion Criteria:

* Uni or bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation

Exclusion Criteria:

* Preceding ocular surgery or trauma
* Recurrent intraocular inflammation of unknown etiology
* Uncontrolled glaucoma
* Uncontrolled systemic or ocular disease
* Blind fellow eye
* Microphthalmus
* Corneal abnormality
* History of uveitis/iritis
* Iris neovascularization
* Pseudoexfoliation
* Proliferative diabetic retinopathy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
IOL rotation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology and Optometry of the Medical University Vienna, Vienna, Vianne, Austria